CLINICAL TRIAL: NCT03845088
Title: Application of Virtual Mandibular Position in Temporomandibular Jont Reconstruction With Costochondral Graft in Children Jaw Deformity.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, shuo chen, Attending Doctor, Peking University
Other Study IDs: schen
Record Dates: First submitted 2018-09-26; First posted 2019-02-19 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Joint Ankylosis; Facial Asymmetry
Keywords: Virtual mandibular position; temporomandibular joint reconstruction; Jaw deformity;Costochondral graft
MeSH Terms: conditions — Temporomandibular ankylosis; Facial Asymmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children TMJA or condyle absence with Jaw Deformity: inclusion criteria: <12 years old; Unilateral temporomandibular joint ankylosis or condyle absence； Temporomandibular joint reconstructed with costochondral graft；
  Interventions: Procedure: temporomandibular jont reconstruction with costochondral transplantation

INTERVENTIONS:
Procedure: temporomandibular jont reconstruction with costochondral transplantation — temporomandibular jont reconstruction with costochondral transplantation guided by virtual mandibular position

SUMMARY:
Hypothesis：Computer-aided design virtual mandibular position is feasible for costochondral graft growing and occlusion stabilizing in the one-stage treatment of children temporomandibular joint ankylosis (TMJA) or condyle absence with jaw deformity.

Methods: The inclusion criteria is children patients younger than 12 years old with unilateral TMJA or condyle absence. A virtual mandibular position is designed preoperatively according to the CT data of jaw and dentition. 3D printed templates and occlusal splints are used to guide the costochondral graft and mandibular position. During surgery, the affected ramus is reconstructed with costochondral grafting under the virtual mandibular position. After surgery, the occlusal splint is fixed to maxilla at least one month, and then, replaced by orthodontic functional appliance to promote downward growth of the maxilla. Occlusion, facial symmetry, costochondral graft growing would be evaluated and analysed until adulthood.

ELIGIBILITY:
Inclusion Criteria:

* <12 years old
* Unilateral temporomandibular joint ankylosis or condyle absence；
* Temporomandibular joint reconstructed with costochondral graft；

Exclusion Criteria:

* Bilateral temporomandibular joint ankylosis or condyle absence
* Combined with systematic disease

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients are surgically treated in the Department of Oral and Maxillofacial Surgery, Peking University School and Hospital of Stomatology, Beijing, China.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bilateral ramus height,chin deviation,maxilla height | preoperation
  Bilateral ramus height,chin deviation,maxilla height in millimeter. These measurements were accomplished by ProPlan 2.0( SynthesProPlan，Materialise，Belgium）
Bilateral ramus height,chin deviation,maxilla height 6 months after operation | 6 months after operation
  Bilateral ramus height,chin deviation,maxilla height in millimeter 6 months after operation. These measurements were accomplished by ProPlan 2.0( SynthesProPlan，Materialise，Belgium）
Bilateral ramus height,chin deviation,maxilla height 12 months after operation. | 12 months after operation
  Bilateral ramus height,chin deviation,maxilla height in millimeter 12 months after operation.These measurements were accomplished by ProPlan 2.0( SynthesProPlan，Materialise，Belgium）

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, PhD, Study Chair — Peking University Hospital of Stomatology
Locations (1):
- Peking University Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data was published 6 months at the end of the trial, through the form of paper publication

REFERENCES:
- [Background] Zhang X, Chen M, Wu Y, Wang B, Yang C. Management of temporomandibular joint ankylosis associated with mandibular asymmetry in infancy. J Craniofac Surg. 2011 Jul;22(4):1316-9. doi: 10.1097/SCS.0b013e31821c9342. PMID 21772189
- [Background] Kaban LB, Perrott DH, Fisher K. A protocol for management of temporomandibular joint ankylosis. J Oral Maxillofac Surg. 1990 Nov;48(11):1145-51; discussion 1152. doi: 10.1016/0278-2391(90)90529-b. PMID 2213309
- [Background] Kaban LB, Bouchard C, Troulis MJ. A protocol for management of temporomandibular joint ankylosis in children. J Oral Maxillofac Surg. 2009 Sep;67(9):1966-78. doi: 10.1016/j.joms.2009.03.071. PMID 19686936
- [Background] Perrott DH, Umeda H, Kaban LB. Costochondral graft construction/reconstruction of the ramus/condyle unit: long-term follow-up. Int J Oral Maxillofac Surg. 1994 Dec;23(6 Pt 1):321-8. doi: 10.1016/s0901-5027(05)80046-3. PMID 7699266
- [Background] Padwa BL, Mulliken JB, Maghen A, Kaban LB. Midfacial growth after costochondral graft construction of the mandibular ramus in hemifacial microsomia. J Oral Maxillofac Surg. 1998 Feb;56(2):122-7; discussion 127-8. doi: 10.1016/s0278-2391(98)90847-3. PMID 9461132
- [Background] Zhu S, Li J, Luo E, Feng G, Ma Y, Hu J. Two-stage treatment protocol for management of temporomandibular joint ankylosis with secondary deformities in adults: our institution's experience. J Oral Maxillofac Surg. 2011 Dec;69(12):e565-72. doi: 10.1016/j.joms.2011.07.025. PMID 22117712
- [Background] Lu C, Huang D, He D, Yang C, Yuan J. Digital occlusal splint for condylar reconstruction in children with temporomandibular joint ankylosis. J Oral Maxillofac Surg. 2014 Aug;72(8):1585-93. doi: 10.1016/j.joms.2013.12.033. Epub 2014 Jan 15. PMID 24613028